CLINICAL TRIAL: NCT02543008
Title: Effect of Physical Activity Following Thoracic Mobilization on Heart Rate Variability and Pressure Pain Threshold in Asymptomatic Subjects: a Randomized Clinical Trial.
Brief Title: Effect of Physical Activity Following Thoracic Mobilization on Heart Rate Variability and Pressure Pain Threshold.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Xavier de Araujo, Pt, Pt, MSc, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUHSPortoAlegre_II
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Asymptomatic individuals
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Physical activity plus thoracic mobilization (Experimental): Subjects randomly allocated to this arm will be submitted to a 10 minutes anaerobic exercise (2 minutes warming up, 5 minutes of 75% to 85% maximal heat rate, 3 minutes slowdown), followed by 5 minutes of passive intervertebral thoracic mobilization (3 sets of 1 minute, grade III, and 1 minute rest between each set).
  Interventions: Procedure: Physical activity plus thoracic mobilization
- Physical activity (Active Comparator): Subjects allocated to this arm will be submitted to the same anaerobic exercise protocol, without the thoracic mobilization.
  Interventions: Procedure: Physical activity
- Placebo (Placebo Comparator): Subjects in this group will be conducted to a placebo thoracic mobilization, without anaerobic exercise protocol. The investigator will apply only a manual contact, to mimic the genuine thoracic mobilization. The same 5 minutes period will be respected, and the same position of therapist and subject.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Physical activity plus thoracic mobilization — Information already included in arm/group descriptions.
  Arms: Physical activity plus thoracic mobilization
Procedure: Physical activity — Information already included in arm/group descriptions.
  Arms: Physical activity
Procedure: Placebo — Information already included in arm/group descriptions.
  Arms: Placebo

SUMMARY:
Comparison of the effects of physical activity (treadmill running) plus thoracic mobilization, physical activity only or a placebo intervention (only manual contact thoracic mobilization), on heart rate variability and pressure pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects
* Sedentary

Exclusion Criteria:

* Spinal pain
* Historic of trauma/surgery to the spine
* Diabetes
* Hypo/hyperthyroidism
* Alcoholic
* Smoker
* Hypertension

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Change from baseline, immediately after, and 15 minutes after the intervention.

SECONDARY OUTCOMES:
Pressure pain threshold | Change from baseline, mimediately after, and 15 minutes after the intervention.
  Digital algometer will be applied to C7 and T4 spinous process, right hand and right tibialis anterior muscle belly

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciencias da Saude, Porto Alegre, Rio Grande do Sul, Brazil